CLINICAL TRIAL: NCT04501939
Title: Cirmtuzumab Consolidation for Treatment of Patients With Detectable CLL on Venetoclax
Acronym: Venetoclax
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Oncternal Therapeutics, Inc (Industry)
Responsible Party: Principal Investigator, Michael Choi, Associate Clin Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191407
Record Dates: First submitted 2020-07-22; First posted 2020-08-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; CLL; cirmtuzumab; venetoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — cirmtuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cirmtuzumab + Venetoclax (Experimental): All patients will receive a minimum of 6 cycles (cycle = 28 days) of therapy with venetoclax and cirmtuzumab during the treatment period. For patients who achieve undetectable minimal residual disease (uMRD) positive after cycle 6, an additional 6 cycles of venetoclax and cirmtuzumab may be administered.
  Interventions: Drug: Cirmtuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Cirmtuzumab — Cycle 1, Day 1 & 15 - 600mg Cycle 2, Day 1 to Cycle 6, Day 1 - 600mg
  Other Names: Zilovertamab
Drug: Venetoclax — Venetoclax 400mg PO daily from cycle 1 day 1 for 6 cycles of 28 days.
  Other Names: VENCLEXTA

SUMMARY:
Single center, open-label, phase 2 study to determine the efficacy of cirmtuzumab consolidation in patients with measurable disease on venetoclax.

DETAILED DESCRIPTION:
This is a phase 2 study to test whether cirmtuzumab in combination with venetoclax given as consolidation therapy can decrease the number of cancer cells that may be left in the bone marrow or in the blood in patients who have been treated with venetoclax for at least one year. Consolidation therapy is given after initial cancer treatment to further reduce the number of cancer cells that may be left in the body. Cirmtuzumab, a monoclonal antibody that inhibits receptor tyrosine kinase like orphan receptor (ROR1) signaling and stemness, may be effective in reducing the risk of disease progression in patients with detectable minimal residual disease (MRD) after treatment with venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Must have detectable CLL/SLL (> 0.01% leukemia cells present)
* Must have received at least 12 months of venetoclax.
* Patients may be receiving venetoclax at the time of screening and study entry.
* Patients who have discontinued venetoclax more than 6 months prior to study entry must still have a disease burden meeting criteria for low risk of TLS (i.e. no lymph node greater than 5 cm in diameter; absolute lymphocyte count less than 25 k/uL)

Exclusion Criteria:

Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

* Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
* Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
* Child class B or C cirrhosis

Treatment with any of the following within 7 days prior to the first dose of cirmtuzumab:

* Steroid therapy for anti-neoplastic intent
* Biologic agent (monoclonal antibody) within 30 days for anti-neoplastic intent.
* Chemotherapy (purine analog or alkylating agent) or target small molecule agent within 14 days or 5 half-lives (whichever is shorter), or has not recovered to less than CTCAE grade 2 clinically significant adverse effect(s)/toxicity(s) of previous therapy.
* CLL therapy, aside from venetoclax.
* History of other malignancy that could affect compliance with the protocol or interpretation of results (example: patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are generally eligible.)
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Cancer response to treatment | 6-24 months
  Percentage of subjects with undetectable measurable residual disease after 6 months of cirmtuzumab + venetoclax treatment.

SECONDARY OUTCOMES:
Frequency of adverse events | 9-15 months
  Number of subjects with treatment-related adverse events as assessed by CTCAE v5.0.
Time to next CLL treatment. | 9-24 months
  Measurement of time of anti-cancer activity

OTHER OUTCOMES:
Change in gene expression in leukemic cells | 9-15 months
  The change in gene expression of leukemia cells by single cell PCR or RNA after treatment with cirmtuzumab, including analysis of archival pre-venetoclax sample, when available.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Heyman, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Koman Family Outpatient Pavilion, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557